CLINICAL TRIAL: NCT06017466
Title: Translation and Implementation of the Dutch VVAS Score in Clinical Practice
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22493VVAS
Record Dates: First submitted 2023-03-15; First posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2022-12

CONDITIONS: Vertigo
Keywords: Vertigo; Epidemiology; Visually Induced Dizziness; Chronic Vertigo
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Intervention Model Description: This will be a prospective interventional study with the Dutch VVAS questionnaire as interventional product.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chronic Vertigo (Experimental): Chronic vertigo patients can be divided into three groups. The first pathway is episodic vertigo (caused by e.g. migraine, Ménière's disease, benign paroxysmal positional vertigo (BPPV)) progressively leading to chronic dizziness. The second pathway is initiated by a single attack of vertigo (e.g. neuritis vestibularis) with some initial recovery but later on residual symptoms. The third pathway is the presence of chronic, slowly progressive, continuous, or unchanging symptoms (e.g. bilateral vestibular failure, CNS disorders). All patient with chronic vertigo (see above) will included.
  Interventions: Diagnostic Test: Visual Vertigo Analogue Scale (VVAS)

INTERVENTIONS:
Diagnostic Test: Visual Vertigo Analogue Scale (VVAS) — The Visual Vertigo Analogue Scale (VVAS) was developed by E. Dannenbaum et al in 2011 to diagnose visual vertigo. It is a nine-item analogue scale in which the subjects can rated the intensity of their symptoms. The symptoms can be categorized as None (0), Mild (0.1-40), Moderate (40.01-70) or Severe (70.01-100). The VVAS is already available in English and French but a Dutch version does not yet exist.

SUMMARY:
The aim of this study is to translate and introduce a cross-cultural adaptation of The Visual Vertigo Analogue Scale (VVAS). E. Dannenbaum et al developed the VVAS in order to diagnose visual vertigo (VV). VV is dizziness caused by visual stimuli such as scrolling through a computer screen or walking through crowds of people or supermarket aisles.

DETAILED DESCRIPTION:
The Visual Vertigo Analogue Scale (VVAS) was developed by E. Dannenbaum et al in 2011 to diagnose visual vertigo. It is a nine-item analogue scale in which the subjects can rate their symptoms' intensity. The symptoms can be categorized as None (0), Mild (0.1-40), Moderate (40.01-70), or Severe (70.01-100). The VVAS is already available in English and French but a Dutch version does not yet exist. In this study, we would like to translate and introduce a cross-cultural adaptation of the VVAS into Dutch for use with vestibular patients in Belgium.

ELIGIBILITY:
Inclusion Criteria:

* All patient with chronic vertigo (>3 years) will included
* Interpretation of the VVAS is be possible
* 18-75 year

Exclusion Criteria:

* Unable to read Dutch
* Single episode of vertigo
* > 75 year
* Minors
* When no interpretation of the VVAS is possible (e.g. too young, dementia)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
vertigo symptoms assessed by the visual analogue scale | 1 year
  Unit of measurement: score from 1 to 10 measurement tool: VVAS questionnaire